CLINICAL TRIAL: NCT06708312
Title: The Effect Of Ears Acupuncture On Fitness Test 12 Minute Running Students Of Medical Faculty UNHAN RI Third Semester
Brief Title: The Effect Of Ears Acupuncture On Fitness Test 12 Minutes Running in Students Of Medical Faculty UNHAN RI
Acronym: sportacup
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Elies Fitriani, MD, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24-09-1517
Record Dates: First submitted 2024-11-24; First posted 2024-11-27 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Sports Physical Therapy; Military Activity; Exercise Overtraining
Keywords: 12 minutes running test; ear acupuncture; sport endurance
MeSH Terms: conditions — Overtraining Syndrome | interventions — Acupuncture, Ear

STUDY DESIGN:
Intervention Model Description: intervention group : ear acupuncture control group : sham ear acupuncture
Who Masked: Participant, Outcomes Assessor
Masking Description: participant blinding by divide into two group randomly and received true ear acupuncture or sham acupuncture randomization were done by research assistant outcome assesed by research assistant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ear acupuncture (Experimental): Placement of pressure needles on the MA-TF1 Shenmen, MA-IC4 Heart and ear points MA-IC4 Sympathetic is carried out 30 minutes before starting the running session. Aseptic and antiseptic measures are carried out with alcohol wipe. Stimulation is carried out at the acupuncture points determined by press for 1 minute, using a press needle measuring 0.22 mm x 15 mm.
  Press the needle removed 15 minutes after the run
  Interventions: Procedure: press needle acupuncture
- sham ear acupuncture (Sham Comparator): Placement of adhesive plaster on the MA-TF1 Shenmen, MA-IC4 Heart ear points and MA-IC4 Sympathetic is carried out 30 minutes before starting the running session. Aseptic and antiseptic measures are carried out with alcohol swab. At acupuncture points, pressure stimulation is not carried out, only rubbing. The adhesive plaster is removed 15 minutes after running.
  Interventions: Procedure: sham press needle acupuncture

INTERVENTIONS:
Procedure: press needle acupuncture — Placement of press needle on the ear acupuncture point : MA-TF1 Shenmen, MA-IC4 Heart, and MA-IC4 Sympathetic
  Other Names: ear acupuncture; earlobe acupuncture
  Arms: ear acupuncture
Procedure: sham press needle acupuncture — Placement of adhesive plaster on the ear acupuncture point : MA-TF1 Shenmen, MA-IC4 Heart, and MA-IC4 Sympathetic
  Arms: sham ear acupuncture

SUMMARY:
The goal of this clinical trial is to study the use of ear acupuncture in 12 minutes running test on third semester of cadets of Medical Faculty, Indonesia Defense University, between intervention and sham group. The outcome measure are heart rate, blood pressure, running distance, intensity and VAS RPE also VAS leg intensity.

DETAILED DESCRIPTION:
Ear acupuncture is a affordable, easy and non-invasive method with good evidence of effectiveness in the scope of physical training. Several previous studies has proven the effectiveness of acupuncture in physical exercise, including helping increases oxygen absorption and reduces lactic acid after exercise, lowering chronic musculoskeletal pain. In reducing pain after physical activity, ear acupuncture has been shown to reduce VAS leg intensity. This shows that ear acupuncture can helps athletes recover after intense training faster. At the Defense University of the Republic of Indonesia (UNHAN RI), Study Program students Bachelor of Medicine (cadet) has both academic demands and military training. The military education demands high stamina and physical fitness. To make sure the cadets are in a fit condition to face daily activities with a busy and numerous schedule physical activity, a physical fitness assessment is carried out at the end of each semester using the 12 run test. By doing this test, principal investigator aims to observe the effect of giving ear press needle acupuncture compare with sham on running 12 minutes in Indonesian Defense University student of medical faculty.

ELIGIBILITY:
Inclusion Criteria:

* Indonesian Defense University Military FK Student Batch 4, Third semester
* Gender male or female, age 18-20 years
* Physically healthy based on the results of medical check-ups in the last 6 months mini medical check up (blood pressure, pulse, saturation, glucose and, Hb check carried out by researchers) as well as being eligible for physical exercise, assessed by PAR-Q questionnaire, history and physical examination
* Willing to follow this research until completion and sign informed consent.
* BMI is normal
* Regularly exercise 5x a week with moderate to heavy intensity categories good physical fitness level
* Do not consume caffeine and high calorie foods high in sugar for 1 hour before the test run

Exclusion Criteria:

* Taking anti-inflammatory drugs (corticosteroids), anti pain (NSAIDS, opioids), muscle relaxants (diazepam, eperisone, etc.) or taking blood thinning drugs (anti-platelet or anti-coagulant drugs).
* Have received any type of acupuncture therapy for some time <7 days before the study.
* History of anti-inflammatory drug treatment in the previous 2 weeks.
* There are tumors, wounds or skin infections, eczema, otitis externa and psoriasis in matchmaking area.
* There was a hypersensitivity reaction to previous acupuncture therapy (allergy metals, severe atopy, keloids, or other skin hypersensitivity).
* Participants had multiple ear piercings.
* Have had surgery on the waist, hip, knee and ankle area before last 1 year.

Ages: 18 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
VO2 max prediction scores | 5, 10, 15 minutes after running sessions
  Reference maximum amount individual capacity in use oxygen during doing activities or exercising, using VO2max prediction scores based on running distance (in meters), then entered into formula (mileage - 504.9 meters)/44.73 and categorized into :
  * Very good
  * OK
  * Enough
  * Less
  * Very less
Blood pressure | 5, 10, 15 minutes after running sessions
  The pressure that occurs on arterial blood vessels when blood is pumped by the heart to be distributed throughout body, units of millimeters of water mercury(mmHg), measured with digital blood pressure meter.
Pulse beat | 5, 10, 15 minutes after running test
  A palpable wave in the arteries when blood is pumped out the heart, reflecting heart rate, counted each the minutes count repetitions (times/min), measurement using digital smart watch
Exercise intensity | after running test, before and after intervention and sham
  The power of deep stimulation exercise, for aerobic exercise heart rate is used. Intensity is categorized in zone, in this study used heavy intensity and maximum 77-100% of HRmax. Measured by Heart rate peak entered into formula Heart rate peak divide into Heart rate maximum x 100%
The Borg rating scale/RPE | 5, 10 , 15 minutes after running test
  The Borg Rating of Perceived Exertion ('Borg' or 'RPE') is a scale used as a indicators to determine energy exerted in a workout with a range 6-20, where 6 means "no exertion at all" and 20 means "maximal exertion."
Modifid borg scale leg fatigue | 5, 10, 15 minutes after running test
  Modified Borg scale to determine size exertion in terms of this is the maximum strength of the leg (inferior extremity) in running with a range of 0-10.0 scale minimum and 10 represents maximum power possible someone tolerates

SECONDARY OUTCOMES:
Adverse event | immediately after and follow up 1 week after running session
  Symptoms reported by patients after receiving press needle acupuncture

CONTACTS AND LOCATIONS:
Overall Officials: KPEK FKUI-RSCM The Health Research Ethic Comittee of Faculty of Medicine, Principal Investigator — Indonesia University
Locations (1):
- Indonesia Defence University, Bogor, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
via the clinicaltrial.org
Supporting Information: Study Protocol, CSR
Time Frame: during this research start november 15th 2024, end november, 15th 2025